CLINICAL TRIAL: NCT04016532
Title: Personalized Dietary Advice After Discharge From Hospital in Geriatrics: Factors Associated With Improved Nutritional Status and Autonomy
Acronym: DIETADOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A03458-47
Record Dates: First submitted 2019-07-03; First posted 2019-07-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-04

CONDITIONS: Undernutrition of Elderly Peopole
Keywords: Elderly peopole; Undernutrition; Acute Geriatric
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient malnourished or at risk of undernutrition (Other): Dietary follow-up at home: 4 visits (D15, D30, D60, D90)
  Interventions: Dietary Supplement: Personalized dietary management at home
- Not undernourished patients (Other): Dietary follow-up at home: 3 visits ( D30,D60, D90)
  Interventions: Dietary Supplement: Personalized dietary management at home

INTERVENTIONS:
Dietary Supplement: Personalized dietary management at home — Personalized dietary management at home to improve nutritional status.
  * Four (J7, J30, J60 and J90 for non-undernutrition patients) or five Home visits (J7, J15, J30 and J90 for undernutrition patients or at risk of undernutrition) by professional dietitians from Saveurs & Vie over a period of 3 months after discharge from the hospital: personalized dietary advice and recipe sheet.
  * There will be no change in medical prescriptions

SUMMARY:
The purpose of this study is to identify the factors associated with the effectiveness of home dietary management in these elderly people returning home (personal home or independent residence) after hospitalization in acute geriatrics.

DETAILED DESCRIPTION:
Patient recruitment will be carried out in the 6 participating hospital centres.

All patients willing to participate, will benefit from an Inclusion Visit (J0): Conducted in hospital in acute geriatric services before discharge from hospital. Verification of inclusion criteria, collection of patient consent by investigator, assignment of patient identification number, declaration of inclusion, and collection by investigator of inclusion data (age, sex, weight, height, appetite, dietary intake scale, risk factors for undernutrition by HAS, albumin, CRP, exit treatment, ADL, IADL and GIR, technical aids for walking, presence of professional and non-professional home workers).

Home visit J7 (30 min to 1 hour): initial dietary assessment, will be carried out between 24 hours and 7 days after discharge from hospital. During this visit, the dietician will perform several measurements (MNA-SF, weight, height, appetite assessment, ingest/24h Consumption of NOCs if prescribed in hospital, Quality of Life, ADL, IADL, acceptance of visit, follow-up of dietary advice and intercurrent medical events).

Home visit J30, J60 (30 min to 1h): Made by the dietician, during these visits will be carried out various measurements and questionnaires: Appetite assessment, weight, ingesta/24h, consumption of NOCs, acceptance of the visit, follow up on dietary advice, compendiums of intercurrent medical events.

Home visit J90 = Final visit. This visit is identical to the initial assessment (J7). Patients who are undernourished or at risk of undernutrition will receive an additional J15 home visit (15 days after discharge from hospital). This visit will be identical to visits J30, J60.

ELIGIBILITY:
Inclusion Criteria:

* Unscheduled hospitalization of at least 4 days in acute geriatrics,
* Direct return to home or independent residence after hospitalization,
* To be domiciled in the Hauts-de-Seine department,
* Good understanding of the French language,
* Beneficiary of a social security scheme,
* Having read the briefing note and having consented to participate in the study by signing a written consent,

Exclusion Criteria:

* Severe cognitive impairment according to DMS-IV criteria,
* Inflammatory syndrome (CRP > 30 mg/l)
* Evolving cancer;
* Chronic respiratory failure,
* Stage IV heart failure
* long-term corticosteroids (> 10 mg/d prednisolone or equivalent),
* Enteral and parenteral nutrition at home,
* Chronic end-stage pathology;
* Inability to walk without human help
* Major person subject to a legal protection measure (guardianship, guardianship and safeguarding of justice)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Screening for undernutrition in geriatric practice according the MNA-SF score (Short-Form Mini-Nutritional Assessment) | 3 months

SECONDARY OUTCOMES:
Assessment of the appetite according the VAS scale "Visual Analog Scale" | 3 months
Assessment of teh degree of autonomy according AGGIR score | Inclusion (0 day)
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 3 months
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | 3 months
Grab force measurement according the dynamometer | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine CHANSIAUX, MD, Study Chair — Geriatric Departement, Rives de Seine hospital
Locations (1):
- Geriactric Departement, Rives de Seine hopsital, Courbevoie, Île-de-France Region, France